CLINICAL TRIAL: NCT02628210
Title: A Prospective, Multi-Center, Non-Randomized Study to Assess Clinical Outcomes Using Interbody Spacers With map3® Cellular Allogeneic Bone Graft in Anterior Lumbar Interbody Fusion or Lateral Lumbar Interbody Fusion
Brief Title: Interbody Spacers With map3® Cellular Allogeneic Bone Graft in Anterior or Lateral Lumbar Interbody Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTI-2014-02
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Spondylosis; Spondylolisthesis; Degenerative Disc Disease
MeSH Terms: conditions — Spondylosis; Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- map3® Cellular Allogeneic Bone Graft (Other): Patients will receive map3® Cellular Allogeneic Bone Graft
  Interventions: Other: map3® Cellular Allogeneic Bone Graft

INTERVENTIONS:
Other: map3® Cellular Allogeneic Bone Graft — Patients will receive map3® Cellular Allogeneic Bone Graft

SUMMARY:
This is a single-arm post-market study in patients requiring lumbar fusion using allograft interbody spacer in conjunction with map3® Cellular Allogeneic Bone Graft in patients with degenerative disc disease (DDD). This cohort study will enroll 80 patients total at up to 10 sites. After subjects have signed an informed consent, the baseline visit and examinations will be completed. Patients will be evaluated at 6 weeks, 3 months, 6 months, 12 months, and 24 month visit after surgery.

DETAILED DESCRIPTION:
Map3 is an allogeneic bone matrix which also contains demineralized cortical cancellous bone and multipotent adult progenitor cells (MAPC). MAPC-based cells are derived from allograft bone marrow, isolated from other cells and cryopreserved. Both the scaffold and cellular constituents are processed from the same donor but are provided in separate containers. Scaffold and cells combined constitute the implant and must be used together. The map3 implant is available in Strips allograft and Chips allograft configurations.

ELIGIBILITY:
Inclusion Criteria:

* is at least 18 - 75 years of age and skeletally mature
* must have symptomatic spondylosis, spondylolisthesis grade I or II, or degenerative disc disease (DDD) at one level from L2-S1 requiring a fusion
* must be a candidate to use an allograft spacer
* must be a candidate for bilateral pedicle screw placement
* must have completed a minimum of six weeks (+/- two to four weeks of bracing) of unsuccessful conservative, non-operative care
* must have discogenic back pain with or without leg pain DDD must be confirmed by MRI or CT scans followed by discography (if necessary)
* must score at least 40 % on the Oswestry Disability Index
* must score 4 or more on a 10 cm Visual Analog Scale for back pain or leg pain
* must be able to comply with the protocol's follow-up schedule
* must understand and sign the informed consent documenT

Exclusion Criteria:

* symptomatic at more than one level
* previous fusion surgery at any lumbar level with or without instrumentation.
* any other bone grafting product other than study product and local autograft bone. e.g. rhBMP2, (recombinant human bone morphogenetic protein 2).
* patients requiring any other interbody fusion device other than an allograft spacer (Bigfoot™, Crossfuse® Advantage). e.g. no PEEK IBF
* more than 50% spondylolisthesis (Myerding grade III or more)
* lumbar scoliosis greater than 11 degrees
* osteoporosis* (T-score of -2.5 or lower), osteomalacia, Paget's disease or --metabolic bone disease.
* spinal tumors
* active arachnoiditis
* fractures of the epiphyseal plate or fractures for which stabilization of the fracture is not possible.
* impaired calcium metabolism
* active infection or surgical site infection
* rheumatoid arthritis or other autoimmune disease that affects bone healing (at the surgeon's discretion)
* chronic steroid use except for chronic inhalers (used steroids for one month within the last 6 months) or any medical condition that requires treatment with drugs known to interfere with bone healing
* use of glucocorticoids > 10 mg/day
* systemic disease such as AIDS, HIV, hepatitis (active), tuberculosis
* morbid obesity defined as body mass index (BMI) >45 or a weight more than 100 lbs. over ideal body weight
* uncontrolled diabetes documented with an Hbg A1C >9 or insulin dependent diabetics
* smokers unless approved by Sponsor, including electronic cigarettes and vaporizers
* within the past two (2) years, psychosocial disorders that would preclude accurate evaluation or has a history of substance abuse any history or active cancer
* pregnancy, or interested in becoming pregnant while participating in the study
* participation in another investigational study within 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in the Oswestry Disability Index (ODI) | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months

SECONDARY OUTCOMES:
Fusion | 6 months, 12 months and 24 months
  Fusion at the operated level, based on
  * Bridging trabecular bone.
  * Less than 3 mm of translational motion.
  * Less than 5 degrees of angular motion.
Changes in Visual Analog Scale (VAS) pain scores. | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
Changes in SF-36 scores. | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
Changes in Lumbar Intervertebral Disc (LID) scores. | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
Changes in medication use | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
Time to return to work | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Chundri, MD, Principal Investigator — Carl & Edyth Lindner Center for Research
Locations (3):
- United States (3):
  - Spine Surgery of Buffalo Niagara, LLC, Niagara Falls, New York
  - AXIS Neurosurgery and Spine of WNY, PLLC, Williamsville, New York
  - Carl & Edyth Lindner Center for Research The Christ Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No